CLINICAL TRIAL: NCT06578039
Title: Single-dose, Phase 1 Clinical Trial to Evaluate the Safety, and Tolerability of Allogeneic Umbilical Cord-derived Mesenchymal Stem Cell Therapy in Patients With Premature Ovarian Insufficiency
Brief Title: Phase 1 Clinical Trial of CordSTEM-ST
Acronym: CBT210-POI_P1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CHABiotech CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBT210-POI_P1
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-08

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Stem cell therapy; allogeneic stem cell; umbilical cord derived mesenchymal stem cell
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group 1 (Low dose CordSTEM-ST) (Experimental): Low dose CordSTEM-ST, 1 (single) administration
  Interventions: Biological: umbilical cord-derived mesenchymal stem cell
- Study Group 2 (High dose CordSTEM-ST) (Experimental): High dose CordSTM-ST, 1 (single) administration
  Interventions: Biological: umbilical cord-derived mesenchymal stem cell

INTERVENTIONS:
Biological: umbilical cord-derived mesenchymal stem cell — allogeneic umbilical cord-derived mesenchymal stem cell
  Other Names: CordSTEM-ST

SUMMARY:
This clinical study will evaluate the safety and tolerability of CordSTEM-ST after administering a single dose in patients with premature ovarian insufficiency (POI), as well as identify the maximum tolerated dose (MTD) and evaluate the potential therapeutic effects.

DETAILED DESCRIPTION:
3 or 6 subjects will be enrolled sequentially by applying the "traditional 3+3 design" to evaluate the dose limiting toxicities (DLTs) for 28 days from the first administration date of the investigational product according to the protocol. A DLT is defined as the occurrence of a grade 3 or higher adverse drug reaction (ADR) according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

First three subjects will be enrolled in Study Group 1 (low dose group) to be evaluated for DLTs up to 28 days after IP administration. If none of three subjects develope DLT, three subjects for Study Group 2 (high dose group) will be recruited. If one out of three subjects in Study Group 1 develop DLT, additional three subjects in Study Group 1 will be enrolled to be evaluated for DLT. If two or more subjects develop DLT in initial three subjects, the study will be terminated.

This study will be followed up by a long-term follow-up study under the separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥ 25 years and < 40 years
* Individuals diagnosed with premature ovarian insufficiency: Individuals who have a follicle stimulating hormone (FSH) level of 40 IU/L or higher in the results of two tests conducted at least 4 weeks apart and are amenorrheic for at least 4 months
* Individuals who voluntarily decide to participate and provide written consent

Exclusion Criteria:

* Individuals diagnosed with primary amenorrhea*

  * No secondary sex characteristics by age 13, Absence of menarche for 5 years after initial breast development, or Absence of menstruation by age 15
* Individuals diagnosed with polycystic ovary syndrome
* Individuals with any other conditions that may affect the result of this study.

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female subjects
Enrollment: 6 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | up to 6 months after the IP administration
  Number of adverse event cases reported
Abnormality cases in lab test results | up to 6 months after the IP administration
  Number of clinically significant abnormalities found in lab test results.
Abnormality cases physical exam results | up to 6 months after the IP administration
  Number of clinically significant abnormalities found in physical exam results
Abnormality cases in vital signs | up to 6 months after the IP administration
  Number of clinically significant abnormalities found in vital signs

SECONDARY OUTCOMES:
Percent change from baseline in blood Follicle Stimulating Hormone (FSH) level | up to 6 months after the IP administration
  blood Follicle Stimulating Hormone (FSH) level measured in mIU/ml
Percent change from baseline in blood Anti-Mullerian Hormone (AMH) level | up to 6 months after the IP administration
  blood Anti-Mullerian Hormone (AMH) level measured in ng/ml
Percent change from baseline blood Estradiaol (E2) level | up to 6 months after the IP administration
  blood Estradiaol (E2) level measured in pg/ml
Percent change from baseline in number of mature follicles | up to 6 months after the IP administration
  number of mature follicles measured in number of follicles
Percent change from baseline in number of antral follicles | up to 6 months after the IP administration
  number of antral follicles measured in number of follicles
Percent change from baseline in endometrial thickness | up to 6 months after the IP administration
  endometrial thickness measured in cm
Status of menstruation resumption | up to 6 months after the IP administration
  Collected by patient interview

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea